CLINICAL TRIAL: NCT02399332
Title: A Collaborative Care Model for Chronic Disease Management in Diabetes - Involvement of Community Pharmacists in Complex Care Plans, a Pilot Study
Brief Title: Involvement of Community Pharmacists in Complex Care Plans for Diabetic Patients, a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Divya Garg, Clinical Assistant Professor, University of Calgary
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB15-0673
Record Dates: First submitted 2015-03-02; First posted 2015-03-26 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community Pharmacist Involvement (Experimental): Patients would have a complex care plan completed by their clinical team, which will involve chronic disease management nurse and the family physician. This complex care plan would also involve discussion with the patient's community pharmacist who would follow-up with the patient monthly and send a report to the patient's physician. Patients would also continue to receive routine care at the clinic.
  The monthly follow-ups with the community pharmacist would involve review of the goals of complex care plan and monitoring clinical targets, medication review and discussing adherence as well as patient education. This follow-up can be completed in person or by telephone. The pharmacist would then send a monthly report to patient's family physician.
  Interventions: Other: Community pharmacist involvement
- Usual care (No Intervention): Patients have a complex care plan completed by their clinical team, which will involve the chronic disease management nurse and the family physician and then receive routine care and follow up. They will receive usual care from their community pharmacist.

INTERVENTIONS:
Other: Community pharmacist involvement — Collaborative involvement of the community pharmacists in formulating and following complex care plans
  Arms: Community Pharmacist Involvement

SUMMARY:
This project is an initiative to bring physicians, nurses, community pharmacists and patients together in collaborative planning in the management of diabetes, which aligns with the collaborative, team based aspects of family medicine as a community based discipline. Alberta funds both physicians and community pharmacists to complete a comprehensive assessment and plan for patients with qualifying medical conditions. Our research hypothesis is that a collaborative approach between healthcare providers involved in delivering care will improve individual patient outcomes with the primary outcome being improved glycemic control. Health care utilization and medication adherence will also be assessed. This project will compare the results of comprehensive annual health care plans implemented over a period of twelve months with or without involvement from community pharmacists. It is hypothesized that involvement of community pharmacists and their collaboration with physicians will lead to improved outcomes.

DETAILED DESCRIPTION:
Research question: Does involvement of a community pharmacist in formulating and following a complex care plan for diabetic patients in conjunction with the patient's clinical team (physician and chronic disease management nurse) improve outcomes including glycemic control, health care utilization and medication adherence.

Hypothesis: Collaborative complex care planning for diabetic patients with the primary care physician, chronic disease management nurse and community pharmacist leads to improvement in patient health outcomes, decreases hospital visits and visits to family physician and emergency room and improves medication adherence.

Aim of the study: The aim of this study is to serve as a pilot in exploring if collaborative care provided by physicians, chronic disease nurse and community pharmacists in formulating and following complex care plans leads to better clinical outcomes when compared to care plans that are formulated and followed in isolation by the physician and chronic disease nurse. This study would be the basis for a future in depth project comparing outcomes of care plans completed in isolation by the pharmacists or physicians with those created in a collaborative environment. Our long-term objectives are improvement in patient outcomes, reduction in health care expenditure as well as preventing duplication and potential discordance of comprehensive care plans.

Methodology

Patients and study design: This is a single centre prospective case control pilot study.

A cohort of 25 eligible diabetic patients at the South Health Campus Family Medicine Teaching Clinic (an outpatient academic family medicine clinic in Calgary, Alberta) will be studied and compared against a group of 25 control diabetic patients. The intervention would be involvement of patient's community pharmacist with their clinical team in formulating the complex care plan and following up with the patient on a monthly basis. The control is a set of patients who have complex care plans completed by their clinical team with no coordination with the pharmacist.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients who have diabetes with HbA1C over target (>7) and who qualify for a complex care plan completion.

Exclusion Criteria:

* Pregnancy
* Unwilling to participate/provide written consent
* Unable or unwilling to participate in planned follow-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in HbA1C from baseline at one year | 1 year

SECONDARY OUTCOMES:
Change in systolic BP from baseline at one year | 1 year
Change in diastolic BP from baseline at one year | 1 year
Change in Low Density Lipoprotein (LDL) from baseline at one year | 1 year
Change in weight from baseline at one year | 1 year
Change in BMI from baseline at one year | 1 year
Change in hospital admissions from baseline at one year | 1 year
Change in family physician visits from baseline at one year | 1 year
Change in emergency room visits from baseline at one year | 1 year
Change in medication adherence from baseline at one year | 1 year